CLINICAL TRIAL: NCT00714155
Title: Outcomes and Patient Satisfaction After Colpocleisis for Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Erin Duecy, MD, University of Rochester
Other Study IDs: 15184
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2011-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: Colpocleisis
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Physical examination, questionnaires, retrospective chart review
  Interventions: Other: Questionnaires, Physical Examination
- 2: Questionnaires, retrospective chart review
  Interventions: Other: Questionnaires, Physical Examination
- 3: Retrospective chart review

INTERVENTIONS:
Other: Questionnaires, Physical Examination — Questionnaires, Physical Examination
  Groups: 1; 2

SUMMARY:
The purpose of this study is to evaluate the long-term success rate of the colpocleisis procedure and its effect on quality of life in women who have this surgery. We want to see if women who have this surgery have problems with recurrent pelvic organ prolapse, urinary incontinence, or bowel problems after the surgery. We also want to see how the surgery affects women's sexuality.

ELIGIBILITY:
Inclusion Criteria:

* women who underwent either total colpectomy with colpocleisis or partial colpectomy with LeFort-type colpocleisis performed by the Urogynecology service between 1/2000 and 12/2007 at Strong Memorial Hospital

Exclusion Criteria:

* women who are not undergone colpocleisis or colpectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Urogynecology clinic
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2006-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Questionnaires | Post-operative

SECONDARY OUTCOMES:
Physical Examination | Post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Erin E. Duecy, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States